CLINICAL TRIAL: NCT04308122
Title: A Randomized Trial of Cervical Orthosis Versus no Orthosis Following Multi-level Posterior Cervical Fusion
Brief Title: Cervical Orthosis Versus no Orthosis Following Multi-level Posterior Cervical Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Christopher Bailey (Other)
Responsible Party: Sponsor-Investigator, Dr. Christopher Bailey, Associate Professor and Staff Physician Department of Surgery, London Health Sciences Centre, The London Spine Centre
Organization: The London Spine Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1 - 22-Apr-2020
Record Dates: First submitted 2020-03-06; First posted 2020-03-13 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Posterior Cervical Spinal Surgery; Myelopathy Cervical; Radiculopathy, Cervical; Spinal Stenosis Cervical; Spondylosis, Cervical
MeSH Terms: conditions — Radiculopathy; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Orthosis (CO) (Active Comparator): Cervical orthosis will be worn at all times for 6 weeks according the standard of care after posterior cervical fusion
  Interventions: Device: Cervical Orthosis (CO)
- No Orthosis (NO) (Experimental): No cervical orthosis will be worn after posterior cervical fusion
  Interventions: Device: No Orthosis

INTERVENTIONS:
Device: Cervical Orthosis (CO) — Immediately following surgery patients in the CO group will be fitted with a Philadelphia collar prior to being transferred to the recovery room. On the patient ward a physiotherapist will fit the patient with a Cervimax/Aspen/Miami J collar which will be worn at all times for 6 weeks according the standard of care.
  Arms: Cervical Orthosis (CO)
Device: No Orthosis — The NO group will have no specific precautions applied to their neck range of motion.
  Arms: No Orthosis (NO)

SUMMARY:
Use of cervical orthosis after instrumented posterior cervical spinal surgery is still widely practiced even though modern fusion techniques likely do not require additional stabilization from an external orthosis. This is a single, centre randomized, non-blinded equivalence trial. Patients undergoing multi-level posterior cervical fusion will be randomized to cervical orthosis (CO group) or no orthosis (NO group). Immediately following surgery patients in the CO group will be fitted with a Philadelphia collar prior to being transferred to the recovery room. On the patient ward a physiotherapist will fit the patient with a Cervimax/Aspen/Miami J collar which will be worn at all times for 6 weeks according the standard of care. The NO group will have no specific precautions applied to their neck range of motion. Outcomes will be assessed prior to surgery, on the second day after surgery, and at 2, 4, 6 and 12 weeks after surgery. The primary outcome will be neck pain score on the numerical rating scale (ranging from 0-10 with higher scores indicating more severe pain) during the first 4 weeks after surgery with an equivalence margin of 2.0 points. Secondary outcomes will be neck disability, general health, treatment satisfaction, pain medication use, adverse events, neck range of motion, time meeting discharge status, and compliance in wearing the collar.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing multi-level (2- or more level), open, posterior cervical fusion which may extent into the second thoracic vertebrae (C1-T2)
2. Able to consent to inclusion in the study
3. 18 years of age and older

Exclusion Criteria:

1. Spinal cord injury
2. Primary cervical spine infection
3. Cervical spine tumor
4. Inability to comprehend patient rated outcome instruments
5. Substance abuse
6. Dementia
7. Psychosis
8. Previous surgery at same level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity | Through study duration to 12 weeks
  numerical rating scale, 0 to 10 with higher scores indicating more severe pain

SECONDARY OUTCOMES:
Neck Disability Index | Through study duration to 12 weeks
  NDI is a self-administered questionnaire with 10 questions. Each question is scored from 0 to 5 for a maximum score of 50 and the score converted to a percentage score. The scale ranges from 0 to 100 with a higher score denoting worse disability.
Arm pain intensity | Through study duration to 12 weeks
  numerical rating scale, 0 to 10 with higher scores indicating more severe pain
General health SF12 | Through study duration to 12 weeks
  is a generic, multidimensional self-report health questionnaireQuestions are categorized into scales for general health, physical functioning, social functioning, role limitation-physical, role limitation-emotional, mental health, energy/fatigue, pain, comparative health. These are summarized into the SF12-physical component summary score (PCS) and mental component summary score (MCS). Scores range from 0 to 100 with higher scores impling better functioning.
Treatment satisfaction (% of patients satisfied) | Through study duration to 12 weeks
  Treatment satisfaction will be assessed by the following question: "Are you satisfied with the results of your spine surgery?" using a 5-category scale as follows: 1) extremely satisfied, 2) somewhat satisfied, 3) Neither satisfied nor dissatisfied, 4) somewhat dissatisfied, 5) extremely dissatisfied.
Time to meet discharge status (days) | day 2
  measured as the number of days it takes to meet all discharge criteria including:
  * Ambulating safely and independently as assessed by the physiotherapist
  * Pain controlled with oral analgesics
  * Minimal wound drainage following drain removal
  * For the CO group only: proficient donning and doffing the CO as assessed by physiotherapy/occupation therapy
Adverse Events rate (%) | Through study duration to 12 weeks
  The Spinal Adverse Events Severity Grading System (SAVES) form will be used to capture intra-operative, peri-operative, and post-operative adverse events and serious adverse events.
Pain medication usage | Through study duration to 12 weeks
  The total dosage of opioids and NSAID for the hospital length of stay will be calculated. The type of medication used (over the counter, NSAID, muscle relaxant, narcotics, anti-depressant, neuroeleptic and other) will be indicated as not taken, as needed, and daily at week 2, 4, 6, and 12 after surgery.
Range of motion | Through study duration to 12 weeks
  Change in cobb angle in flexion-extension xrays and a goniometer to measure flexion-extension and rotation
Compliance with wearing the collar (collar group only) | Through study duration to 12 weeks
  Patients will be asked they used the collar as prescribed. If not, they will be asked if they wore the collar at all, and if yes for how many hours per day. Compliance will be defined as prescribed, irregular or aborted. Patients will be compliant if they wear the collar for> 20 hours per day.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bailey, Principal Investigator — London Health Science Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandes R, Thornley P, Urquhart J, Alahmari A, Alenezi N, Kelly S, Rasoulinejad P, Singh S, Siddiqi F, Gurr K, Bailey C. Cervical orthosis does not improve postoperative pain following posterior cervical fusion: a randomized controlled trial. Eur Spine J. 2024 Oct;33(10):4002-4011. doi: 10.1007/s00586-024-08456-7. Epub 2024 Aug 21. PMID 39167110